CLINICAL TRIAL: NCT04671511
Title: Sentinel Node Biopsy and Targeted Axillary Dissection in Node-Positive Breast Cancer Patients With Clinically Negative Axilla
Brief Title: Targeted Axillary Dissection (TAD) in Early-stage Node Positive Breast Cancer
Acronym: TADEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Quebec Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Jean-Francois Boileau, MD, MSc, FRCSC, Surgical Oncologist, Associate Professor Surgery and Oncology, McGill University, Director JGH Breast Clinical Trials Group, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-05-2021-2605
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female; Early-stage Breast Cancer; Lymph Node Metastases; Axillary Metastases; Sentinel Lymph Node
Keywords: breast cancer; targeted axillary dissection; sentinel lymph node biopsy; clinically negative axilla; metastatic axillary lymph nodes
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Axillary Dissection (Experimental): Ultrasound of the axilla preoperative. Clipped biopsy proven positive node. I125 radioactive seed before surgery. Sentinel node biopsy using Tc99 +/- blue dye. Targeted Axillary Node Dissection performed at surgery
  Interventions: Procedure: Targeted Axillary Dissection; Diagnostic Test: Ultrasound of the axilla

INTERVENTIONS:
Procedure: Targeted Axillary Dissection — Sentinel Node Biopsy (SNB; using Tc99 +/- Blue dye) + Radioactive Seed Localisation (RSL) of clipped node using I125 seed = Targeted Axillary Dissection (TAD)
Diagnostic Test: Ultrasound of the axilla — Prospectively recorded preoperative ultrasound of the axilla. Number of suspicious nodes recorded. Biopsy and clipping of the positive node.

SUMMARY:
RATIONALE: It is now standard for most breast cancer patients with 1-2 positive sentinel nodes to avoid completion node dissection when eligibility criteria from the American College of Surgeons Oncology Group (ACOSOG) Z0011 trial are met. The National Comprehensive Cancer Network (NCCN) recently proposed to extend this indication to patients that present with biopsy proven node positive disease if only 1 or 2 suspicious nodes are found on imaging, these positive nodes are not palpable clinically, and the other eligibility criteria from the Z0011 study are otherwise met. However, this recommendation is based on an expert consensus and no study has yet confirmed the optimal method to stage the axilla in this patient population.

PURPOSE: Evaluate the technical success rate and accuracy of sentinel node biopsy (SNB) and the potential benefits of clipping and removing the biopsy proven node using radioactive seed localisation (RSL) (SNB+RSL = Targeted Axillary Dissection (TAD)) in patients with biopsy proven positive nodes, limited nodal disease in imaging and clinically negative axillary examination.

DETAILED DESCRIPTION:
This is a prospective multicenter study. Patients with T1-2 Breast cancer and clinically negative axilla on palpation, 1-2 suspicious nodes on ultrasound, and a biopsy proven positive node (by core biopsy of fine needle aspiration) will have a radioactive seed (I125) placed in their clipped node before surgery. At the time of surgery, patients that are scheduled for breast conserving surgery or mastectomy will have sentinel node biopsy (SNB) using radioactive dye (Tc99) +/- blue dye as well as retrieval of the clipped node using radioactive seed localisation (RSL). Removal of the I125 radioactive seed in the clipped node will be performed before the Tc99 counts are performed to prevent "shine through" and biased measurements. Imaging of the surgical specimen will confirm retrieval of the clipped node. Prospectively recorded information on pre-operative axillary imaging, characteristics of the retrieved nodes in the operating room and detailed pathological analysis of each corresponding node will be performed. Completion node dissection (CND) is not mandatory in this study but recommended if the clipped positive node is not retrieved, if 4 nodes or more are positive or if 3 nodes are positive in the absence of axillary radiation. The benefits of adding RSL to SNB and the benefits of adding SNB to RSL staging of the axilla will be evaluated in this study and will help to better define the value of using TAD in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years old.
* Participants with a clinical T1 or T2 invasive ductal or lobular breast carcinoma, regardless of estrogen/progesterone/human epidermal growth factor receptor 2 (HER2) receptor status.
* Participants with clinical (on palpation) N0 and up to two suspicious lymph nodes on axillary ultrasound.
* Participant with biopsy-proven positive axillary disease made by core needle biopsy or fine-needle aspiration.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status less than 2.
* Participants must understand, accept, and have signed the approved consent form.

Exclusion Criteria:

* Participant with previous ipsilateral axillary surgery, including sentinel lymph node biopsy.
* Participants with distant metastases.
* Participants that have had previous radiotherapy to the axillary nodes.
* Participants who received neoadjuvant therapy.
* If the injection of blue dye is planned, patients with hypersensitivity or allergy to isosulfan blue, patent blue, methylene blue or radiocolloid dye.
* Participants who are unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in recommended completion node dissection rate (CND) with the use of Targeted Axillary Dissection (TAD) vs. Sentinel Node Biopsy (SNB) alone. | 1 month
  Recommended completion node dissection rate (CND) = false negative rate (FNR) + technical failure rate (TFR).
  TAD CND (TAD FNR + TAD TFR) vs. SNB CND (SNB FNR + SNB TFR)

SECONDARY OUTCOMES:
Identification rate of patients with three or more positive nodes using only radioactive seed localisation (RSL) vs. Targeted Axillary Dissection (TAD) | 1 month
  Evaluate if the addition of SNB to RSL improves the ability to identify patients with 3+ positive nodes that do not otherwise meet the ACOSOG Z0011 criteria and require further regional axillary therapy
False negative rate (FNR) of Targeted Axillary Dissection (TAD) | 1 month
  Percentage of patients with successful removal of at least one node (using this method) where at least one positive node was not retrieved (using this method)
Technical failure rate (TFR) of Targeted Axillary Dissection (TAD) | 1 month
  Percentage of patients with unsuccessful removal of at least one node using this method, including the clipped node
False negative rate (FNR) of Radioactive Seed Localisation (RSL) | 1 month
  Percentage of patients with successful removal of at least one node (using this method) where at least one positive node was not retrieved (using this method)
Technical failure rate (TFR) of Radioactive Seed Localisation (RSL) | 1 month
  Percentage of patients with unsuccessful removal of at least one node using this method, including the clipped node
False negative rate (FNR) of Sentinel Node Biopsy (SNB) | 1 month
  Percentage of patients with successful removal of at least one node (using this method) where at least one positive node was not retrieved (using this method)
Technical failure rate (TFR) of Sentinel Node Biopsy (SNB) | 1 month
  Percentage of patients with unsuccessful removal of at least one node using this method (clipped node or not)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Boileau, MD,MSc,FRCSC, Study Chair — Jewish General Hospital; Léamarie Meloche-Dumas, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Erica Patocskai, MD, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (3):
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Giuliano AE, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Hunt KK, Morrow M, Ballman K. Locoregional recurrence after sentinel lymph node dissection with or without axillary dissection in patients with sentinel lymph node metastases: the American College of Surgeons Oncology Group Z0011 randomized trial. Ann Surg. 2010 Sep;252(3):426-32; discussion 432-3. doi: 10.1097/SLA.0b013e3181f08f32. PMID 20739842
- [Background] Mansel RE, Fallowfield L, Kissin M, Goyal A, Newcombe RG, Dixon JM, Yiangou C, Horgan K, Bundred N, Monypenny I, England D, Sibbering M, Abdullah TI, Barr L, Chetty U, Sinnett DH, Fleissig A, Clarke D, Ell PJ. Randomized multicenter trial of sentinel node biopsy versus standard axillary treatment in operable breast cancer: the ALMANAC Trial. J Natl Cancer Inst. 2006 May 3;98(9):599-609. doi: 10.1093/jnci/djj158. PMID 16670385
- [Background] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Costantino JP, Ashikaga T, Weaver DL, Mamounas EP, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Wolmark N. Sentinel-lymph-node resection compared with conventional axillary-lymph-node dissection in clinically node-negative patients with breast cancer: overall survival findings from the NSABP B-32 randomised phase 3 trial. Lancet Oncol. 2010 Oct;11(10):927-33. doi: 10.1016/S1470-2045(10)70207-2. PMID 20863759
- [Background] Giuliano AE, Ballman KV, McCall L, Beitsch PD, Brennan MB, Kelemen PR, Ollila DW, Hansen NM, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Morrow M. Effect of Axillary Dissection vs No Axillary Dissection on 10-Year Overall Survival Among Women With Invasive Breast Cancer and Sentinel Node Metastasis: The ACOSOG Z0011 (Alliance) Randomized Clinical Trial. JAMA. 2017 Sep 12;318(10):918-926. doi: 10.1001/jama.2017.11470. PMID 28898379
- [Background] Benson AB, Venook AP, Al-Hawary MM, Arain MA, Chen YJ, Ciombor KK, Cohen SA, Cooper HS, Deming DA, Garrido-Laguna I, Grem JL, Hoffe SE, Hubbard J, Hunt S, Kamel A, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Nurkin S, Overman MJ, Parikh A, Patel H, Pedersen KS, Saltz LB, Schneider C, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Johnson-Chilla A, Gregory KM, Gurski LA. Small Bowel Adenocarcinoma, Version 1.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Sep 1;17(9):1109-1133. doi: 10.6004/jnccn.2019.0043. PMID 31487687
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Background] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Background] Boileau JF, Poirier B, Basik M, Holloway CM, Gaboury L, Sideris L, Meterissian S, Arnaout A, Brackstone M, McCready DR, Karp SE, Trop I, Lisbona A, Wright FC, Younan RJ, Provencher L, Patocskai E, Omeroglu A, Robidoux A. Sentinel node biopsy after neoadjuvant chemotherapy in biopsy-proven node-positive breast cancer: the SN FNAC study. J Clin Oncol. 2015 Jan 20;33(3):258-64. doi: 10.1200/JCO.2014.55.7827. Epub 2014 Dec 1. PMID 25452445
- [Background] Classe JM, Loaec C, Gimbergues P, Alran S, de Lara CT, Dupre PF, Rouzier R, Faure C, Paillocher N, Chauvet MP, Houvenaeghel G, Gutowski M, De Blay P, Verhaeghe JL, Barranger E, Lefebvre C, Ngo C, Ferron G, Palpacuer C, Campion L. Sentinel lymph node biopsy without axillary lymphadenectomy after neoadjuvant chemotherapy is accurate and safe for selected patients: the GANEA 2 study. Breast Cancer Res Treat. 2019 Jan;173(2):343-352. doi: 10.1007/s10549-018-5004-7. Epub 2018 Oct 20. PMID 30343457
- [Background] Caudle AS, Yang WT, Krishnamurthy S, Mittendorf EA, Black DM, Gilcrease MZ, Bedrosian I, Hobbs BP, DeSnyder SM, Hwang RF, Adrada BE, Shaitelman SF, Chavez-MacGregor M, Smith BD, Candelaria RP, Babiera GV, Dogan BE, Santiago L, Hunt KK, Kuerer HM. Improved Axillary Evaluation Following Neoadjuvant Therapy for Patients With Node-Positive Breast Cancer Using Selective Evaluation of Clipped Nodes: Implementation of Targeted Axillary Dissection. J Clin Oncol. 2016 Apr 1;34(10):1072-8. doi: 10.1200/JCO.2015.64.0094. Epub 2016 Jan 25. PMID 26811528
- [Background] Caudle AS, Yang WT, Mittendorf EA, Black DM, Hwang R, Hobbs B, Hunt KK, Krishnamurthy S, Kuerer HM. Selective surgical localization of axillary lymph nodes containing metastases in patients with breast cancer: a prospective feasibility trial. JAMA Surg. 2015 Feb;150(2):137-43. doi: 10.1001/jamasurg.2014.1086. PMID 25517573